CLINICAL TRIAL: NCT06766045
Title: Comparison of Ultrasound with Fluoroscopy to Assess Diaphragmatic Paralysis After Congenital Heart Disease Surgery
Acronym: USG vs Fluoro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Responsible Party: Principal Investigator, Sisca Natalia Siagian, Physician of Pediatric Cardiology and Congenital Heart Disease, Principal Investigator, National Cardiovascular Center Harapan Kita Hospital Indonesia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DP.04.03/KEP162/EC087/2023
Record Dates: First submitted 2024-12-27; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Diaphragmatic Paralysis
Keywords: Diaphragmatic ultrasound; Fluoroscopy; Diaphragmatic paralysis; Congenital heart disease surgery
MeSH Terms: conditions — Respiratory Paralysis | interventions — Fluoroscopy

STUDY DESIGN:
Masking Description: Two different clinicians performed fluoroscopy and diaphragmatic ultrasound without knowing the results of the other tests.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Assessment of Diaphragmatic Paralysis after Congenital Heart Disease Surgery (Experimental): The included patients who were suspected of diaphragmatic paralysis based on clinical symptoms and X-ray examination would first undergo fluoroscopy test, continued by ultrasound examination less than 24 hours apart. The patients were weaned off from mechanical ventilation (spontaneous breathing) and switched to minimal mechanical ventilation support (CPAP/P SIMV) before the examination. The examination and data collection were performed by two different operators: diaphragmatic ultrasound by pediatric intencivist and fluoroscopy test by pediatric cardiologist.
  Interventions: Diagnostic Test: Diaphragmatic Ultrasound; Diagnostic Test: Fluoroscopy

INTERVENTIONS:
Diagnostic Test: Diaphragmatic Ultrasound — Diaphragmatic ultrasound was performed bedside in the ICU with supine position. Diaphragmatic thickness was measured by placing the ultrasound on 8th-10th intercostal space between anterior and mid-axillary line with marker at 12 o'clock. B-mode ultrasound was used to measure the distance between thoracic and abdominal diaphragm which resulted in the diaphragmatic thickness at inspiration (DTi) and diaphragmatic thickness at expiration (DTe).
  The ultrasound was then placed on the subcostal area between anterior and mid-axillary line with marker at 12 o'clock to observe the diaphragmatic motion on each side. Measurement of diaphragmatic excursion as well as recording and evaluation of diaphragmatic sliding and motion were performed during both inspiration and expiration using M-mode.
Diagnostic Test: Fluoroscopy — Fluoroscopy test was conducted in cathlab with supine position and anteroposterior (AP) projection for at least 5 breathing cycles. The fluoroscopy recording was then expertised and interpreted by the pediatric cardiologist in charge.

SUMMARY:
Diaphragmatic paralysis after congenital heart disease (CHD) surgery can increase patient mortality and morbidity, especially for the vulnerable pediatric patient. Establishing a diagnosis of this disorder is key for making follow-up decisions such as diaphragm plication. Fluoroscopy as the gold standard has limitations in assessing diaphragmatic paralysis after CHD surgery Objective: To compare diaphragmatic ultrasound with fluoroscopy as the diagnostic method for diaphragmatic paralysis after CHD surgery.

DETAILED DESCRIPTION:
Diaphragmatic paralysis is a common cause of delayed recovery and morbidity after cardiovascular surgery which accounts for 64% of all causes of phrenic nerve lesions. Similarly, congenital heart disease surgery is commonly associated with phrenic nerve injury resulting in diaphragmatic dysfunction in pediatric patients with an incidence of 0.3-5.4%. The phrenic nerve can be injured through various mechanisms such as hypothermia due to ice cold slush for myocardial protection, dissection near the pedicle area of the internal thoracic artery, dissection or conduction of heat along the path or area of the phrenic nerve, etc. Diaphragmatic paralysis is usually transient and not clinically significant in adult, but it is a serious and life-threatening complication that causes respiratory distress in pediatric patient.

Various diagnostic techniques can be used to assess diaphragmatic paralysis such as chest X-ray, fluoroscopy, computed tomography (CT), dynamic magnetic resonance imaging (MRI), and electromyography. The fluoroscopy test has been the method of choice to diagnose diaphragmatic paralysis as it is relatively easy to perform. Earlier studies diagnosed unilateral diaphragmatic paralysis by evaluating the dynamic motion of the diaphragm using fluoroscopy. However, there are several disadvantages of fluoroscopy tests such as requiring cooperation from the patient, requiring the patient in an upright position, the difficulty in transporting patients from the ICU to the fluoroscopy room or cath lab, especially in unstable patients who may deteriorate, the cumulative burden of exposure to radiation, and the relatively high costs.

Diaphragmatic ultrasound (two-dimensional combined with M-mode) is a fast, simple, cheap, accurate, non-radiation noninvasive study that is widely available and increasingly used both in clinical setting and researches. Bedside ultrasound can be used for immobilized or intensive care patients. The simpler procedure helps assessing diaphragmatic paralysis in pediatric patients. The combination of B-mode and M-mode in ultrasound can quantitatively assess the distance and amplitude of diaphragm motion on both sides so that it may provide objective quantification. Therefore, this study was conducted to compare diaphragmatic ultrasound with fluoroscopy as the diagnostic method of diaphragmatic paralysis after congenital heart disease surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had congenital heart disease (CHD) surgery in National Cardiovascular Center Harapan Kita (NCCHK)
* Suspected of diaphragmatic paralysis based on clinical symptoms and X-ray examination.

The conditions indicating diaphragmatic paralysis in patients after CHD surgery were mechanical ventilation dependence, increased respiratory effort and reduced peripheral oxygen saturation when breathing spontaneously, recurrent respiratory tract infection, and chest X-ray showing right hemidiaphragm >2 cm higher than left diaphragm or left diaphragm at the same level or higher than right diaphragm

Exclusion Criteria:

* Patients who could not achieve oxygen saturation targets with the help of minimal pressure support such as continuous positive airway pressure (CPAP) or pressure support intermittent mandatory ventilation (P SIMV)
* Refusal from the patient/family to be included in the study
* Past medical history of diaphragmatic disorder.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) | through study completion, an average of 2 years

SECONDARY OUTCOMES:
Incidence of Diaphragmatic Paralysis after congenital heart disease surgery | through study completion, an average of 2 years
Distress Events during Fluoroscopy and Ultrasound test | through study completion, an average of 2 years
  During both procedures, patients' conditions were documented to monitor any distress event. Distress event was positive if the patients' conditions met one of these criteria: (1) increased heart rate > 90th percentile based on age according to Pediatric Advanced Life Support (PALS), (2) decreased heart rate < -90th percentile based on age according to PALS, (3) cardiac arrest, (4) life-threatening arrhythmia, (5) decreased peripheral oxygen saturation >20% from baseline/preprocedure, (6) increased body temperature >38oC, and (7) partial or generalized seizure.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cardiovascular Center Harapan Kita, Jakarta, DKI Jakarta, Indonesia